CLINICAL TRIAL: NCT05566145
Title: Evaluation of a Back-to-home Support Program for Hospitalized Patients for Heart Failure
Acronym: PRADO_IC2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PRADO St Jo
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients included in the PRADO program: Patients hospitalized for global heart failure or left ventricular insufficiency in the Cardiology department of the GHPSJ between January 2016 and September 2018, included in the support program for Return To Home for Heart Failure (PRADO)
- Patients not included in the PRADO program: Patients hospitalized for global heart failure or left ventricular insufficiency in the Cardiology department of the GHPSJ between January 2016 and September 2018, not included in the Return A DOmicile support program for Heart Failure (PRADO)

SUMMARY:
The prevalence of heart failure is very high worldwide is between 1 and 2% in developed countries.

The French Federation of Cardiology estimates that a million people are affected in France. Each year in France, there are nearly 70,000 deaths linked to heart failure, and more than 150,000 hospitalizations with an average cumulative duration per year of 12.7 days, figures which show the extent of the phenomenon. Heart failure is therefore a common pathology, which constitutes an important public health issue. It requires rigorous monitoring and early adaptation of treatments to avoid repeated hospitalizations. Studies show that following hospitalization for heart failure, all-cause re-hospitalization rates rise to 18% within 30 days. In 2019, the rate of re-hospitalization at 1 year is 30%, half of which in the following 3 months. The prognosis is grim with 20 to 30% of deaths within the year.

The European Society of Cardiology recommends that the patient be integrated into a care path coordinated by the general practitioner; and a consultation with his general practitioner in the week after hospitalization and his cardiologist within two weeks. The CPAM (Caisse Primaire d'Assurance Maladie) has set up since 2013 the PRADO-IC program (Program for Return to Home Hospital for Heart Failure). This program must be in place before discharge from hospital. A health insurance advisor comes to meet the patient, declared eligible for PRADO by the hospital medical team, to present the offer and collect his approval before discharge. He then contacts the attending physician and organizes his return home. A follow-up book is given to the patient to allow better transmission of information between town and hospital.

A specially trained nurse visits the patient's home every week. The duration of PRADO support varies according to the NYHA stage of severity. It provides therapeutic education with reinforcement of hygieno-dietetic rules, warning signs, checks compliance with treatments and the necessary biological monitoring and must alert the attending physician in the event of aggravation.

The objectives of this program are: to preserve the quality of life and the autonomy of patients, to support the reduction of the length of stay in hospital, to strengthen the quality of care in town around the attending physician, improve the efficiency of recourse to hospitalization by reserving the heaviest structures for the patients who need them most.

DETAILED DESCRIPTION:
The prevalence of heart failure is very high worldwide: according to the European Society of Cardiology, it is between 1 and 2% in developed countries.

The French Federation of Cardiology estimates that a million people are affected in France. This prevalence increases sharply with age, reaching 15% of people aged 85 and over.

Each year in France, there are nearly 70,000 deaths linked to heart failure, and more than 150,000 hospitalizations with an average cumulative duration per year of 12.7 days, figures which show the extent of the phenomenon. In addition, the aging of the population and the explosion of cardiovascular risk factors suggest that the impact of heart failure will be greater in the future.

Heart failure is therefore a common pathology, which constitutes an important public health issue. It requires rigorous monitoring and early adaptation of treatments to avoid repeated hospitalizations. Studies show that following hospitalization for heart failure, all-cause re-hospitalization rates rise to 18% within 30 days. According to a report from the Caisse Primaire d'Assurance Maladie (CPAM) in 2019, the rate of re-hospitalization at 1 year is 30%, half of which in the following 3 months. The prognosis is grim with 20 to 30% of deaths within the year.

The European Society of Cardiology recommends that the patient be integrated into a care path coordinated by the general practitioner; and a consultation with his general practitioner in the week after hospitalization and his cardiologist within two weeks. But general practitioners deplore a lack of coordination between city and hospital with difficulties in taking care of their patient following hospitalization. According to the CPAM report, only 30% of re-hospitalized patients had contact with a cardiologist before their readmission, and 15% of patients had no contact with the health care system within 2 months of followed their hospitalization.

It is in this need to improve monitoring that the CPAM has set up since 2013 the PRADO-IC program (Support Program for Return to Home Hospital for Heart Failure). This program must be in place before discharge from hospital. A health insurance advisor comes to meet the patient, declared eligible for PRADO by the hospital medical team, to present the offer and collect his approval before discharge. He then contacts the attending physician and organizes his return home. A follow-up book is given to the patient to allow better transmission of information between town and hospital.

A specially trained nurse (internet training) visits the patient's home every week. The duration of PRADO support varies according to the NYHA stage of severity: a patient in NYHA stage I or II benefits from home support for a period of 2 months, and 6 months for NYHA stages III and IV. It should make it possible to monitor the constants: blood pressure, pulse, and weight. It provides therapeutic education with reinforcement of hygieno-dietetic rules (low sodium diet), warning signs (orthopnea, cough, dyspnea), checks compliance with treatments and the necessary biological monitoring and must alert the attending physician in the event of aggravation.

The objectives of this program are: to preserve the quality of life and the autonomy of patients, to support the reduction of the length of stay in hospital, to strengthen the quality of care in town around the attending physician, improve the efficiency of recourse to hospitalization by reserving the heaviest structures for the patients who need them most.

The main objective of this study is to evaluate the impact of the PRADO program on morbidity and mortality in a retrospective cohort of heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

For the PRADO Cohort

* Male or female whose age is ≥ 18 years
* Patient hospitalized for heart failure in the GHPSJ Cardiology Department between September 2016 and December 2018 included in the PRADO program
* Patient affiliated to a CNAM IDF social security scheme (general scheme a priori)
* Patient understanding the research issues

For the control cohort

* Male or female whose age is ≥ 18 years
* Patient hospitalized for congestive heart failure (ICD 10 code I500) or left ventricular failure (ICD 10 code I501) in the GHPSJ Cardiology department between September 2016 and December 2018
* Patient affiliated to a social security scheme CNAM IDF
* Patient discharged to home
* Not included in the PRADO program
* Patient who understands the research issues

Exclusion Criteria:

* Patient transferred to another establishment or service (surgery, follow-up care, EHPAD...)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient at the end of life whose vital status is engaged
* Patient who objects to the use of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for global heart failure or left ventricular failure in the Cardiology department of the GHPSJ between January 2016 and September 2018.
Sampling Method: Non-Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of the PRADO program on morbidity and mortality | Year 1
  This outcome corresponds to the combined rate of all-cause mortality and all-cause re-hospitalization at 1 year, wherever it occurred.

SECONDARY OUTCOMES:
Mortality at 1 year | Year 1
  This outcome corresponds to the mortality at 1 year.
First re-hospitalization | Year 1
  This outcome corresponds to the delay until the first re-hospitalization during the year.
Time limit for the use of professionals | Year 1
  This outcome corresponds to the time to first consultation with a general practitioner in town.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ABASSADE, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Gheorghiade M, Vaduganathan M, Fonarow GC, Bonow RO. Rehospitalization for heart failure: problems and perspectives. J Am Coll Cardiol. 2013 Jan 29;61(4):391-403. doi: 10.1016/j.jacc.2012.09.038. Epub 2012 Dec 5. PMID 23219302
- [Background] Albert NM, Barnason S, Deswal A, Hernandez A, Kociol R, Lee E, Paul S, Ryan CJ, White-Williams C; American Heart Association Complex Cardiovascular Patient and Family Care Committee of the Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Transitions of care in heart failure: a scientific statement from the American Heart Association. Circ Heart Fail. 2015 Mar;8(2):384-409. doi: 10.1161/HHF.0000000000000006. Epub 2015 Jan 20. PMID 25604605